CLINICAL TRIAL: NCT03986346
Title: The Vascularity Changes of Scars With Receiving Pulsed Dye Laser
Brief Title: The Vascularity Changes of Scars With Laser Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Chinese University of Hong Kong (Other); Southwest Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20190402002
Record Dates: First submitted 2019-05-24; First posted 2019-06-14 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2019-05

CONDITIONS: Hypertrophic Scar
Keywords: hypertrophic scar; pulsed dye laser
MeSH Terms: conditions — Cicatrix, Hypertrophic | interventions — Lasers, Dye

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser group (Experimental): Participants in this group receive pulsed dye laser to treat the scar.
  Interventions: Device: pulsed dye laser; Other: standardized care
- Control group (Active Comparator): Participants in this group receive standardized care.
  Interventions: Other: standardized care

INTERVENTIONS:
Device: pulsed dye laser — The scar will receive PDL 585 nm using a 7 mm spot size. First treatment will be within 1 year post injury.
  Arms: Laser group
Other: standardized care — the scar will receive standardized care such as scar massage.

SUMMARY:
The purpose of this study is to explore the effects of pulsed dye laser on managing scar vascularity and thickness.

DETAILED DESCRIPTION:
The pulsed dye laser is increasingly used in clinical settings to manage scars and shows promising outcomes.The pulsed dye laser targets at micro-vascular structures in scar tissues. This study aims to explore the vascularity changes in scars with pulsed dye laser during the scar formation process.

ELIGIBILITY:
Inclusion Criteria:

* scars caused by burn injury or related trauma;
* wound healing days over 3 weeks;
* days post injury less than 1 year;
* ability and willingness to comply with all the treatment and assessment procedures.

Exclusion Criteria:

* history of steroid injection or graft surgery;
* history of keloid scarring;
* open wound or active infection;
* conditions that affect wound healing, such as diabetes mellitus.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
scar erythema | 3 months
  Dermoscopy captures the scar photo and measures degrees of scar erythema.
scar blood flow | 3 months
  Ultrasound measures blood flow in scar tissues
scar thickness | 3 months
  Ultrasound measures scar thickness.

SECONDARY OUTCOMES:
patient and observer scar assessment scale (POSAS) | 3 months
  The POSAS measures scar vascularity, pigmentation, pigmentation, thickness, relief, pliability and surface area. Every parameter ranges from 1 to 10, and higher score indicates worse scar performance in that parameter. The total score of POSAS is calculated by summing all the parameters' scores.

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Li-tsang, Principal Investigator — The Hong Kong Polytechnic University
Locations (2):
- Southwest Hospital, Chongqing, China
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deng H, Li-Tsang CWP. Measurement of vascularity in the scar: A systematic review. Burns. 2019 Sep;45(6):1253-1265. doi: 10.1016/j.burns.2018.10.026. Epub 2018 Dec 10. PMID 30545695